CLINICAL TRIAL: NCT06171763
Title: The Multi-stakeholder Assessment of Economic and Managerial Determinants and Impacts of Telemedicine: a Comparison Between a Tele-homecare Solution and Traditional Care Models.
Brief Title: The Multi-stakeholder Assessment of Economic and Managerial Determinants and Impacts of Telemedicine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Buzzi Children's Hospital (Other)
Responsible Party: Principal Investigator, Valeria Calcaterra, Clinical Professor, Buzzi Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0033846
Record Dates: First submitted 2023-11-28; First posted 2023-12-15 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Telemedicine
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehome care (Experimental): For patients/caregivers assigned to the tele-homecare group, before discharge, instruction on the use of the TytoCareTM system was provided by healthcare personnel trained in the use of the system. Subsequently, each patient give the device they used until the scheduled post-discharge clinical assessment. A parent/caregiver was invited to participate for each pediatric patient.
  Every 24 hours, the patient was assessed remotely in synchronous teleconsultation by medical staff; during tele-visit, the physician performed the complete routine procedure, including medical history and physical examination with user friendly medical device and completed the data collection sheet.
  At 72 hours after discharge, an in-person clinical assessment was scheduled for outcome evaluation. In particular, during the visit, the complete resolution of the disease state was assessed through the post-discharge objective examination.
  Interventions: Other: Telemedicine
- Standard care (No Intervention): Patients remained hospitalized for the continuation of the treatment. Every 24 hours, the patient was assessed in person by medical staff; the traditional physical examination involved assessment of the clinical parameters using standard equipment such as a digital thermometer, conventional stethoscope, and otoscope and completed the same data collection sheet.
  After 72 hours of hospital observation, an in-person clinical examination was conducted to evaluate the outcome. In particular, during the visit, the complete resolution of the disease state was assessed through the post-discharge objective examination.

INTERVENTIONS:
Other: Telemedicine — The telehomecare solution involves an early discharge with continued home monitoring through the use of telemedicine utilizing an user-friendly mobile. Additionally, there were a clinical reassessment in person 72 hours after discharge to evaluate the outcomes and results of the intervention.
  Arms: Telehome care

SUMMARY:
The study aims to conduct a comprehensive evaluation involving multiple stakeholders to assess the factors influencing and the consequences of telehomecare in comparison to traditional care models. The integration of technology into the healthcare sector necessitates significant changes in care of patients, organizational structures, production processes, organizational responsibilities, and the management of service delivery processes.

The delivery of telemedicine services through integrated devices represents a method of service production that demands active involvement from patients or, in the case of pediatric patients, their caregivers. This collaborative process of patient engagement in healthcare services is referred to as "co-production." In this research, telehomecare will be examined as an illustrative instance of co-producing healthcare services.

Co-production implies that the inputs into a production process are contributed not only by the organization producing a good or service but also by the users. In the case study, co-production occurs through the interaction between patients/caregivers and professionals during telehealth visits for device-mediated monitoring activities. Throughout the televisit, patients/caregivers play a crucial role in collecting and sharing the necessary parameters with professionals using the device, thereby serving as essential actors in the care process.

The investigators explored the impact of a transitional care program, utilizing an user-friendly mobile medical device, to support an early discharges in a pediatric setting. Clinical outcome and economic advantages are considered. This study will contribute to implement knowledge on the role of telemedicine on HaH healthcare in pediatrics.

DETAILED DESCRIPTION:
This is a single-center, two-arm, randomized, open-label, parallel-group study that was conducted at Buzzi Children's Hospital, a hospital in a metropolis located in Milan (Italy). The different arms consisted of an experimental group with an early discharge adopting telehomecare and a standard care group with in-person physical care until the end of hospitalization.

ELIGIBILITY:
Inclusion criteria:

* Age: 0-18 years.
* Gender: Both males and females
* Patients: Hospitalized at the end of treatment.
* Stable Vital Signs (heart rate, respiratory rate, oxygen saturation)
* Stable/Improving/Resolved biochemical Tests.
* Absence of Fever
* Consent/Assent: Willingness to participate with appropriate consent or assent based on age.
* Proximity to Domicile: Residence within a maximum distance of 45 minutes.
* Adequate Home Facilities.
* Language Proficiency: Adequate knowledge of the Italian language.
* Possession of Compatible Device

Exclusion criteria:

* Refusal to Participate
* Vital Signs Instability
* Presence of Fever
* Deteriorating biochemical Test Results
* Residence More Than 45 Minutes Away
* Inadequate Home Facilities
* Language Barrier
* Lack of a Compatible Device
* Not owning a device with an operating system suitable for supporting the Tytocare app.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Early discharge utilizing an user-friendly mobile medical device | 12 months
  Considering in-person visit as the standard care procedure, the primary objective of this study is to obtain concordance with complete resolution of the disease from in-person physical care, without re-admission to the hospital. The investigators expect non-readmission in a minimum of 90 % of cases.
  Outcome measure: count and percentage of patients readmitted to the hospital after early discharge

SECONDARY OUTCOMES:
Length of stay | 12 months
  To record a lower length of stay in interventional group compared to standard care group Outcome measure: days of hospitalization
Economic impact | 12 months
  To compare costs of hospitalization between interventional group compared to standard care group Outcome measure: direct and indirect costs (in euros)

CONTACTS AND LOCATIONS:
Locations (1):
- Buzzi Children's Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No